CLINICAL TRIAL: NCT02557542
Title: Pilot Randomised Controlled Trial Evaluating the Potential Benefit of a One Stop Vein Clinic (OSVeC)
Brief Title: Pilot RCT Evaluating a One Stop Vein Clinic
Acronym: OSVeC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very poor recruitment
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14/LO/1295
Record Dates: First submitted 2015-08-26; First posted 2015-09-23 (Estimated); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Varicose Veins
Keywords: Varicose Veins; One Stop Clinic
MeSH Terms: conditions — Varicose Veins | interventions — Radiofrequency Ablation; Polidocanol; Sodium Tetradecyl Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- One Stop Vein Clinic (Experimental): Patients randomised to this group will be invited to the One Stop Vein Clinic, offering same day diagnosis and treatment
  Interventions: Other: One Stop Vein Clinic; Device: Radiofrequency ablation; Device: Endovenous laser ablation; Drug: Foam sclerotherapy (Polidocanol or Sodium Tetradecyl Sulphate)
- Normal Care Pathway (Active Comparator): Patients randomised to this group will be invited to the Normal Care Pathway
  Interventions: Other: One Stop Vein Clinic; Device: Radiofrequency ablation; Device: Endovenous laser ablation; Drug: Foam sclerotherapy (Polidocanol or Sodium Tetradecyl Sulphate)

INTERVENTIONS:
Other: One Stop Vein Clinic — Same day diagnosis and treatment
Device: Radiofrequency ablation — Venous ablation
Device: Endovenous laser ablation — Venous ablation
Drug: Foam sclerotherapy (Polidocanol or Sodium Tetradecyl Sulphate) — Venous ablation

SUMMARY:
A pilot randomised controlled trial looking at the setting up of a one stop vein clinic for the treatment of varicose veins and assessing the quality-adjusted life years at 3 months of patients This will be a pilot study which is designed to provide enough information for a potentially larger multicentre randomised controlled study.

DETAILED DESCRIPTION:
OBJECTIVES

* Primary Objective

  o Measure the quality-adjusted life years (QALY) gained at 3 months (using EuroQoL's EQ-5D) & AVVQ by patients randomised to treatment in the One Stop Vein Clinic with patients randomised to treatment in the normal care pathway
* Secondary Objective

  * Patient satisfaction with the service provided using the Picker patient experience questionnaire both post-operatively and at the 3 months follow-up (One Stop Vein Clinic versus Normal Care Pathway)
  * Measure and compare the quality of life scores using CIVIQ at 0 and 3 months in patients randomised to treatment in the One Stop Vein Clinic with patients randomised to the Normal Care Pathway
  * Record the time from referral to treatment (RTT)
  * Assess the cost-effectiveness of the One Stop Vein clinic compared to the normal care pathway
  * Record the time to return to normal activities and to work
  * Assess the estimated societal costs

BACKGROUND Varicose veins are very common conditions, affecting approximately 25% of the population. Over 35,000 varicose vein procedures are currently carried out in the UK. However, with the new 2013 NICE guidelines, the Department of Health has estimated that this is set to increase to 50,000 per year. Waiting for varicose vein interventions has been shown to be detrimental to the severity of the condition and the quality of life of patients. Progression of varicose veins can also lead to complications such as leg ulcerations and can be costly to the health service. Over the past decade, new endovenous techniques have been introduced and these are felt to be cost-effective, especially, when performed in an outpatient or 'office-based' setting. At present, patients referred to the Vascular unit for consideration of management of their varicose veins have to attend the outpatient clinic at least twice prior to be listed for their procedure.

At present, patients referred to the Vascular Outpatient Clinics for consideration for varicose vein management have an initial appointment where the severity of the venous insufficiency is assessed clinically and, subsequently, have a venous Duplex scan to evaluate the extent and cause of any venous incompetence. If any treatable lesion is found, they are then added to the waiting list to come for the eventual varicose vein procedure. This means, they have to attend at least two outpatient appointments and attend another appointment for their venous scans, before actually attending for their varicose vein procedure. Waiting for varicose vein interventions has been shown to lead to worsening of their conditions both clinically and radiologically. In addition, the quality of life of patients waiting for elective surgery is adversely affected.

In order to evaluate patients' ideas and expectations with respect to the provision of varicose vein service in the investigator's unit, they conducted a survey of patients attending the Vascular Outpatient Clinic between March and June 2014. One hundred and six patients completed the anonymous questionnaire. Most were females (62.4%) with a mean age of 51 ± 15 years. More than 90% of patients stated that the waiting time between a Vascular appointment and a venous scan should be no more than 1 month and 85% of patients believed varicose vein procedures should be received within 1 month of their Vascular clinic appointment. Ninety percent of patients were agreeable to attend a 'one-stop' vein clinic offering same day diagnosis and treatment. Patients were generally accepting of the fact that most procedures would be carried out under local anaesthetic (89%).

Hence, it appears that patients in this unit have a preference for a one stop clinic. This concept is not new and has been piloted in other specialities with good success - a one-stop carpal tunnel clinic as well as a one stop cataract clinic was shown to be feasible with good patient satisfaction. Both laparoscopic and open inguinal hernia repairs, where patients received a general anaesthetic, have been carried out successfully using a one stop model offering same day diagnosis and treatment. There is currently already a 'see and treat' service for skin lumps operating at many NHS Trusts and there is already a one stop carpal tunnel service being provided at the Imperial College NHS Trust. It would appear that these one stop clinics have the advantage of reducing the number of unnecessary hospital visits as well as possibly leading to cost savings to the health service.

As a result, the investigators intend to evaluate the one stop model within their own varicose vein service. They will assess the feasibility of having a one-stop vein clinic, where patients will be assessed, have their venous Duplex scans and, depending on the lesions shown, have their venous treatment on the same day.

The hypothetical benefits of such a stratagem are an improvement in patient satisfaction, a reduction in the number of appointments, the abolition of any waiting times as well as cost savings to the health savings.

METHODS GP referrals will be screened and patients meeting the inclusion criteria will be invited to take part in the trial .

They will be sent an information pack containing:

1. Information leaflet about the trial
2. Information about varicose veins, their treatments and a telephone number as a helpline
3. The Aberdeen Varicose Vein Questionnaire (AVVQ), the Chronic Venous Disease Quality of Life Questionnaire (CIVIQ) and EuroQoL's quality of life questionnaire (EQ-5D)
4. Consent form to participate in the study

Patients agreeing to be part of the trial will be consented and randomised either to:

1. The One Stop Vein Clinic (offering same day diagnosis and treatment); or
2. The normal care pathway

Once patients indicate their consent to participate, their General Practitioners (GP) will be sent a letter informing them of the patient's participation in this study.

Patients declining to partake in the randomised part of the study, but agreeable to complete study questionnaires while continuing down the normal care pathway, will also be consented. Further information will be provided to them when they attend for their clinic appointment and the consenting process will take place when they attend for their subsequent procedure

One Stop Vein Clinic Pathway

Patients attending the One Stop Vein Clinic will be reviewed by the Vascular Surgeon, who will confirm the patient's consent in the trial, then assess the degree of venous disease and fill in the Clinical-Etiology-Anatomy-Pathophysiology (CEAP) classification and Varicose Clinical Severity Score (VCSS). If the patient's symptoms are deemed secondary to venous disease, they will be sent to have a Duplex scan to confirm the presence of the venous disease. The results will be reviewed by the Vascular Surgeons, and if the patients are suitable for endovenous ablation +/- avulsions or UGFS, they will be informed of the findings of the scan and proposed treatment. If they are happy to go ahead with the proposed intervention, they will be consented and transferred to the waiting area to wait for their intervention. If, however, they decline same day treatment, they will be put onto the conventional care pathway.

Another Vascular Surgeon will be carrying out the interventions in an 'office-based' environment under local anaesthetic. Once done, the patients will be asked to fill the Picker patient experience questionnaire. They will subsequently be discharged, similar to current practice, and will be given a diary card to fill for when they return to their normal activities and work.

Three (3) months post-operatively, they will be asked to fill the AVVQ, CIVIQ, EQ-5D and Picker patient experience questionnaires once more. This will be done by sending them the questionnaires by post.

The Normal Care Pathway (NCP)

In the normal care pathway, patients referred by their GP are seen in the outpatient clinic and, if their symptoms are suggestive of varicose vein disease, they are sent to have a venous duplex scan. This usually happens on a different day. Afterwards, they are seen back in the clinic (again on a different day) and, if the scan result suggests venous incompetence amenable to day case treatment, they are added to the waiting list. The eventual procedure takes place some time later (within 18 weeks from referral to treatment). After their procedure, they will be asked to fill a Picker patient experience questionnaire. On discharge, they will be given a diary card to fill for when they return to their normal activities and work.

At 3 months post intervention, patients randomised to the normal care pathway will be sent the QoL questionnaires again and asked to fill the AVVQ, CIVIQ, EQ-5D and Picker patient experience questionnaires. As there will be an inherent delay in the NCP pathway, the time from randomisation cannot be used as many patients will not have received their interventional treatment by then.

Inclusion and Exclusion Criteria

The inclusion criteria are:

1. Adults over the age of 18 years
2. Unilateral lower limb symptoms suggestive of venous disease on the referral letter

The exclusion criteria are:

1. Recurrent varicose veins
2. Known arterial disease or ABPI<0.8
3. Current deep vein thrombosis
4. Patients who withdraw their consent
5. Inability to complete the questionnaire or attend follow up appointments
6. Currently enrolled in other venous study

PATIENT SELECTION This is a pilot randomised controlled study and patients will be selected following screening of the GP referral letter.

CONSENT As part of the consenting process, patients will be given three options.

1. Patients wishing to attend the One Stop Vein Clinic and participate in the study will be asked to indicate their consent by signing a consent form and filling in a reply slip. Patients will be randomised either to the One Stop Vein Clinic group or to the Normal Care Pathway (NCP) group.
2. Patients not wishing to attend the One Stop Vein Clinic and participate in the study will be asked to indicate this by filling in a reply slip. They will instead attend the normal care pathway. They will, however, be asked, if agreeable to complete the QoL and Picker patient experience forms.
3. Patients declining either the trial or simple service evaluation will be offered the NCP.

TREATMENT ALLOCATION Treatment received will depend on the findings on the venous Duplex scan. All treatments are minimally invasive with endovenous ablation procedures (either radio-frequency ablation, endovenous laser ablation or mechano-chemical ablation), avulsions or ultrasound-guided foam sclerotherapy. All procedures will be carried out under local anaesthetic and patients will be discharged home later that day, as is the current standard of care.

MEASUREMENT OF OUTCOMES

Primary Outcome

• Measure the quality-adjusted life years (QALY) gained at 3 months (by patients randomised to treatment in the One Stop Vein Clinic with patients randomised to treatment in the Normal Care Pathway)

Secondary Outcome

* Patient satisfaction with the service provided using the Picker patient experience questionnaire both post-operatively and at the 3 months follow-up (One Stop Vein Clinic versus Normal Care Pathway)
* Measure and compare the quality of life scores using EQ-5D, AVVQ and CIVIQ at 0 and 3 months in patients randomised to treatment in the One Stop Vein Clinic with patients randomised to the Normal Care Pathway
* Time from referral to treatment
* Assess the cost-effectiveness of the One Stop Vein clinic compared to the normal care pathway
* Record the time to return to normal activities and to work
* Assess the estimated societal costs

STUDY DURATION & SAMPLE SIZE Following screening of their GP referral letter, patients with varicose vein disease will be invited to participate in the study. It is estimated that 12-14 patients will be invited on a weekly basis to participate in the study following screening. Out of those, only 8 patients is expected to agree to be randomised to the One Stop Vein Clinic or Normal Care Pathway. If the clinic is held weekly, approximately 416 patients could be recruited over the course of the year (8 patients X 52 weeks).

Statistical analysis suggests that the sample size of 208 patients per group would be able to power a potential phase 3 multicentre randomised controlled trial. Compared to a previous study conducted in the investigators' unit which involved 317 patients in total and looked at different quality of life scores and their responsiveness11, the coefficient of variation (ratio of standard deviation to mean) was found to increase at the follow-up period and to vary among the different scores used. With a larger sample size as in this pilot study, this variability would be reduced and result in a smaller coefficient of variation when looking at the follow-up scores. Hopefully, this will enable us to identify the QoL score with the least variability and use it as the primary outcome measure in a future Phase 3 study. A primary outcome measure with little variability would provide us with enough information to estimate an adequate sample size for any future randomised controlled trials.

For example, with a sample size of 208 patients and coefficient of variation of 0.5, a 15% reduction in the geometric mean (a measure of central tendency, similar to median) would be required compared to 25% from the Shepherd et al. study. With power at 85%, this would allow us to determine an adequate sample size.

Participants will be followed-up post-procedure for 3 months, including for patients randomised to the Normal Care Pathway (with potentially longer waiting time from referral to treatment). This means that the study period will be about 18 months. With 3 months for study start-up and 3 months to write the study up, the study will last for 24 months. Approximately 1,000 patients undergo varicose vein procedures at the Imperial College NHS Trust every year.

COST BENEFIT OF PROJECT The hypothesis is that along with improved patient satisfaction and improved waiting times for outpatient appointment, there will be cost savings derived from the One Stop Vein Clinic. On average, 1,000 patients are treated every year in the Imperial College NHS Trust and the cost of an outpatient attendance is approximately £93. Savings could be made if patients are seen and treated at their first appointment rather than having to attend another two appointments.

The potential cost saving is estimated to be in the order of £186,000 annually (£93 x 1,000 X 2).

Estimated societal costs. Data will be collected on time off from work and carer's duties (child/relative/friend). Additionally, data on income, cost of attending clinic and impact on family and colleagues will be assessed to estimate the societal cost of the two pathways.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 years
* Unilateral lower limb symptoms suggestive of venous disease on the referral letter

Exclusion Criteria:

* Recurrent varicose veins
* Known arterial disease or ABPI<0.8
* Current deep vein thrombosis
* Patients who withdraw their consent
* Inability to complete the questionnaire or attend follow up appointments
* Currently enrolled in other venous study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Charing Cross Hospital, Imperial College London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | One Stop Vein Clinic | Normal Care Pathway
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Poor recruitment | 3 | 0

BASELINE CHARACTERISTICS:
Population: No patient recruited to normal care pathway
Groups:
- Total: Total of all reporting groups
Arm/Group | One Stop Vein Clinic | Normal Care Pathway | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Continuous [Median (Full Range); unit: years] | 60 [28 to 76] |  | 60 [28 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 0 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life Using EuroQoL EQ-5D
Description: Quality of life using the EuroQoL EQ-5D scale which is a generic quality of life score. Minimum score = -0.073 (worse) and maximum score is 1.0 (best).
Time Frame: 3 months
Population: Data was not collected from any participants at 3 months due to early study termination
Arm/Group | One Stop Vein Clinic | Normal Care Pathway
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction using a patient satisfaction questionnaire. Minimum score = 0 and maximum score = 10.
Time Frame: 3 months
Population: Data was not collected from any participants at 3 months due to early study termination
Arm/Group | One Stop Vein Clinic | Normal Care Pathway
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Generic Quality of Life Scores Using EQ-5D Questionnaire
Description: EuroQoL's EQ-5D instrument -> Measures health-related quality of life (minimum score = -0.073 (worst); maximum score = 1.0 (best)).
Time Frame: 3 months
Population: Data was not collected from any participants at 3 months due to early study termination
Arm/Group | One Stop Vein Clinic | Normal Care Pathway
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Specific Quality of Life Scores Using AVVQ
Description: Aberdeen Varicose veins Questionnaire -> disease-specific quality of life questionnaire (Minimum score = 0 (best); Maximum score = 100 (worst)).
Time Frame: 3 months
Population: Data was not collected from any participants at 3 months due to early study termination
Arm/Group | One Stop Vein Clinic | Normal Care Pathway
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time From Referral to Treatment
Description: Time from referral from GP to intervention. Number of patients treated within 18 weeks. Minimum = 0 and maximum = number of patients recruited in the study.
Time Frame: 18 weeks
Population: Data was not collected from any participants at 3 months due to early study termination
Arm/Group | One Stop Vein Clinic | Normal Care Pathway
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Measure the Cost of the One Stop Vein Clinic Compared to the Normal Care Pathway
Description: Cost of treating patients through the normal referral pathways compared to treating them on the intervention pathway
Time Frame: 3 months
Population: Data was not collected from any participants at 3 months due to early study termination
Arm/Group | One Stop Vein Clinic | Normal Care Pathway
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Report the Time to Return to Normal Activities and to Work
Description: Time to return to normal activities or to work for patients on the normal referral pathway and intervention group.
Time Frame: 1 month
Population: Data was not collected from any participants due to early study termination
Arm/Group | One Stop Vein Clinic | Normal Care Pathway
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Measure the Societal Costs of the One Stop Vein Clinic
Description: Comparing societal costs with the normal referral pathway compared to the new intervention pathway
Time Frame: 3 months
Population: Data was not collected from any participants at 3 months due to early study termination
Arm/Group | One Stop Vein Clinic | Normal Care Pathway
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Poor recruitment, therefore, study terminated early
Arm/Group | One Stop Vein Clinic | Normal Care Pathway
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-03-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT02557542/Prot_000.pdf